CLINICAL TRIAL: NCT07211152
Title: A Phase Ⅲ, Randomized, Double-blind, Positive Controlled Clinical Trial to Evaluate the Immunogenicity and Safety of an Influenza Vaccine (Split Virion), Inactivated, Quadrivalent in Pregnant Women
Brief Title: Influenza Vaccine (Split Virion), Inactivated, Quadrivalent in Pregnant Women
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-QINF-3006
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Influenza
Keywords: pregnant women
MeSH Terms: conditions — Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Participants will receive one dose of vaccine (0.5 mL) of Sinovac QIV
  Interventions: Biological: Participants will receive one dose of vaccine (0.5 mL) of Sinovac QIV
- Control Group (Active Comparator): Participants will receive one dose of vaccine (0.5 mL) of Vaxigrip QIV
  Interventions: Biological: Vaxigrip QIV

INTERVENTIONS:
Biological: Participants will receive one dose of vaccine (0.5 mL) of Sinovac QIV — Participants will receive one dose of vaccine (0.5 mL) of Sinovac QIV
  Arms: Test Group
Biological: Vaxigrip QIV — Participants will receive one dose of vaccine (0.5 mL) of Vaxigrip QIV
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, positive controlled phase Ⅲ clinical trial to assess the immunogenicity and safety of Sinovac QIV in pregnant women. A total of 150 healthy pregnant women aged 18~39 years at 20 to 32 weeks of pregnancy will be enrolled. All participants will be randomized to test group and control group in a ratio of 2:1 and receive one dose of vaccine (0.5 mL) of Sinovac QIV or Vaxigrip QIV, respectively.

Blood samples will be collected from participants prior to vaccination and 28 days after vaccination. Moreover, to evaluate trans-placental antibodies, blood samples at the end of the gestation period (delivery) and the cord blood sample will be collected, if applicable.

For safety assessment, any immediate adverse events within 30 minutes, solicited local and systemic adverse events within 7 days and unsolicited adverse events within 28 days will be collected. Serious adverse events will be collected within 8 weeks after delivery. Pregnancy and birth outcomes will be collected as well.

DETAILED DESCRIPTION:
This is a randomized, double-blind, positive controlled phase Ⅲ clinical trial to assess the immunogenicity and safety of Sinovac QIV in pregnant women. A total of 150 healthy pregnant women aged 18~39 years at 20 to 32 weeks of pregnancy will be enrolled. Written informed consent form (ICF) will be obtained from participants before enrollment. All participants will be randomized to test group and control group in a ratio of 2:1 and receive one dose of vaccine (0.5 mL) of Sinovac QIV or Vaxigrip QIV, respectively.

For immunogenicity assessment, blood samples will be collected from participants prior to vaccination and 28 days after vaccination. Moreover, to evaluate trans-placental antibodies, blood samples at the end of the gestation period (delivery) and the cord blood sample will be collected, if applicable.

For safety assessment, any immediate adverse events within 30 minutes after vaccine administration, solicited local and systemic adverse events within 7 days and unsolicited adverse events within 28 days will be collected. Serious adverse events will be collected within 8 weeks after delivery. Pregnancy and birth outcomes will be collected by medical record review from enrollment through hospital discharge following delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged 18 to 39 years in good health or medically stable.
2. Gestational age of 20 to 32 weeks, based on last menstrual period, early or late ultrasound dating.
3. The participant was tested negative for HIV, Syphilis, Hepatitis B, Hepatitis C infection according to medical records or rapid tests.
4. Participants should provide verifiable identification.
5. Participants are able to understand and sign the informed consent form voluntarily;
6. Participants are willing and able to adhere to visit schedules and all study requirements.

Exclusion Criteria:

1. Receipt of any seasonal influenza vaccine within 6 months prior to enrollment, or plans to receive other influenza vaccines during the study;
2. Participants with previous or concurrent dangerous pregnancy complications such as gestational diabetes mellitus (GDM), pregnant induced hypertension, preeclampsia and known uterine anomaly;
3. History of preterm delivery, or spontaneous abortion;
4. Known fetal congenital anomaly, e.g. genetic abnormality or major congenital malformation based on antenatal ultrasound;
5. Signs or symptoms of active preterm labor, defined as regular uterine contractions with cervical change (dilation/effacement);
6. History of Guillain-Barré syndrome within 6 weeks of a prior dose of any influenza vaccine;
7. Received any vaccine in the 4 weeks prior to study vaccination, or plans to receive any vaccine within 4 weeks after study vaccination;
8. Serious allergic reaction or other serious adverse reaction to any influenza vaccines or their components;
9. Autoimmune diseases, immunodeficiency, any immunosuppressant within 6 months prior to vaccination (≥ 20mg/day prednisone or equivalent, but corticosteroid spray therapy for allergic rhinitis and surface corticosteroid therapy for acute non-concurrent dermatitis are permitted) or cytotoxic therapy, or plans for such treatment during the study;
10. Diagnosed abnormal coagulation function (e.g., coagulation factor deficiency, coagulation disorders, or platelet abnormalities), or obvious bruising following venipuncture;
11. Significant chronic diseases that, in the judgement of the investigator, might interfere with the study (may include, but are not limited to cardiovascular disease, liver or kidney disorders, HIV infection or malignant tumor);
12. Current or history of severe neurological diseases (such as epilepsy, convulsions or seizures) or psychiatric disorders, or family history of psychiatric disorders;
13. Acute diseases or acute stage of chronic diseases within 7 days prior to vaccination;
14. Receipt of blood, blood-derived products or immunoglobulins within 3 months prior to vaccination or plans for such treatment in the study;
15. Alcoholism or history of drug abuse;
16. Receipt of other investigational drugs/vaccines within 30 days prior to enrollment, or plan to receive investigational drugs/vaccines during the study period;
17. Fever on vaccination day, with axillary temperature ≥ 37.3°C pre-vaccination;
18. Any other factors which are unsuitable for participation in the clinical trial as judged by the investigator.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of hemagglutination inhibition (HI) antibodies against each antigen 28 days after vaccination. | 28 days after vaccination
  SCR 28 days after vaccination.
The seroprotection rates (SPRs) of hemagglutination inhibition (HI) antibodies against each antigen 28 days after vaccination. | 28 days after vaccination
  SPR 28 days after vaccination.
The geometric mean titers (GMTs) of hemagglutination inhibition (HI) antibodies against each antigen 28 days after vaccination. | 28 days after vaccination
  GMT 28 days after vaccination.
The geometric mean increase (GMI) of hemagglutination inhibition (HI) antibodies against each antigen 28 days after vaccination. | 28 days after vaccination
  GMI 28 days after vaccination.
Incidence of adverse reactions within 28 days after vaccination | 28 days after vaccination
  Incidence of adverse reactions within 28 days after vaccination

SECONDARY OUTCOMES:
The maternal seroconversion rates (SCRs) of HI antibodies against each antigen at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  SCRs at the end of gestation period
The maternal seroprotection rates (SPRs) of HI antibodies against each antigen at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  SPRs at the end of gestation period
The maternal geometric mean titers (GMTs) of HI antibodies against each antigen at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  GMTs at the end of gestation period
The maternal geometric mean increase (GMI) of HI antibodies against each antigen at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  GMI at the end of gestation period
The SPR of HI antibodies against each antigen in the umbilical cord blood at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  SPR in the umbilical cord blood at the end of gestation period
The GMT of HI antibodies against each antigen in the umbilical cord blood at the end of gestation period | at the end of gestation period (date of delivery, estimated to be 4-17 weeks after randomization)
  GMT in the umbilical cord blood at the end of gestation period
Incidence of adverse reactions within 7 days after vaccination. | 7 days after vaccination
  Adverse reactions within 7 days after vaccination.
Incidence of serious adverse events within 8 weeks after delivery. | 8 weeks after delivery
  serious adverse events within 8 weeks after delivery.
Incidence of pregnancy and birth outcomes | 8 weeks after delivery
  pregnancy and birth outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Philippines (2):
  - Health Cube Medical Clinics, Mandaluyong, National Capital Region
  - University of the Philippines - Philippine General Hospital (UP-PGH), Manila, National Capital Region

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) may be shared on reasonable request.